CLINICAL TRIAL: NCT05057130
Title: Neoadjuvant Three-component Chemotherapy Based on a Combination of Doxorubicin, Cisplatin and Methotrexate in Patients Aged 24-40 Years With Primary Bone Tumors to Increase the Response Rate Compared With Two-component Chemotherapy
Brief Title: Neoadjuvant Combination of Doxorubicin, Cisplatin and Methotrexate in Patients Aged 24-40 Years With Primary Bone Tumors
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAP2021-7-2
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Osteosarcoma; Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Sarcoma; Sarcoma of Bone
Keywords: Bone sarcoma
MeSH Terms: conditions — Osteosarcoma; Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Sarcoma; Bone Neoplasms | interventions — Doxorubicin; Cisplatin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Three-component chemotherapy (Experimental): Doxorubicin 25 mg / m2 IV on days 1-3, Cisplatin 120 mg / m2 IV on day 1 against the background of hyperhydration. G-CSF support from 4 to 13 days. Methotrexate 12 g / m2 at 28 and 35 days IV with leucovorin 60 mg / m2 in the first 5 days after each administration of methotrexate. The interval between cycles is 42 days
  Interventions: Drug: Doxorubicin, Cisplatin, Methotrexate
- Two-component chemotherapy (Active Comparator): Doxorubicin 25 mg / m2 IV on days 1-3, Cisplatin 120 mg / m2 IV on day 1 against the background of hyperhydration. G-CSF support from 4 to 13 days. The interval between cycles is 28 days
  Interventions: Drug: Doxorubicin, Cisplatin

INTERVENTIONS:
Drug: Doxorubicin, Cisplatin, Methotrexate — IV
  Other Names: MAP
  Arms: Three-component chemotherapy
Drug: Doxorubicin, Cisplatin — IV
  Other Names: AP
  Arms: Two-component chemotherapy

SUMMARY:
Two cycles of neoadjuvant three-component chemotherapy according to the MAP prototoc: Doxorubicin 25 mg / m2 IV on days 1-3, Cisplatin 120 mg / m2 IV on day 1 against the background of hyperhydration. G-CSF support from 4 to 13 days. Methotrexate 12 g / m2 at 28 and 35 days IV with leucovorin 60 mg / m2 in the first 5 days after each administration of methotrexate. The interval between cycles is 42 days.

The advantage of this regimen is to use the three-component chemotherapy regimen, which should increase the degree of tumor necrosis and increase the rate of tumor response to treatment, which will further improve the disease prognosis. Currently, the use of such treatment for adult patients (over 24 years old) is controversial. Since it is believed that the elimination of methotrexate in adult patients is more delayed than in patients under 24 years old, and can lead to serious adverse events (SAE). However, the use of modern standard methods of hemodialysis makes it possible to avoid SAE.

DETAILED DESCRIPTION:
The role of methotrexate in neoadjuvant chemotherapy for bone tumors is a topic for debate. However, the benefits of methotrexate have been confirmed in at least one phase II study showing better results with high doses of methotrexate in the context of triple chemotherapy. Moreover, many studies have shown a correlation between peak serum methotrexate levels, tumor response to chemotherapy, and treatment outcome. Thus, it is possible that the negative results of the effectiveness of methotrexate have been compromised due to the administration of insufficient doses or incorrect administration of the drug. The optimal regimen of methotrexate administration has not been established. However, the control group in the EURAMOS-1 study of the American Osteosarcoma Research Group (AOST) is considered as the standard. The main practical problem with the use of triple chemotherapy in a group of patients aged 24 and older is that the slow clearance of methotrexate can delay the administration of the next cycle of doxorubicin-cisplatin, thereby reducing the dose intensity and adversely affecting the outcome. Currently, there are both isolated clinical cases and observations of a small number of included patients. The use of three-component neoadjuvant chemotherapy for primary bone tumors will improve the rate of response to treatment, reduce the frequency of recurenses and disease progression.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of primary bone tumor (osteosarcoma)

Age from 24 to 40 years

Operable process, possibility of performing resection R0-R1

ECOG performance score 0 or 1

Normal renal function (estimated creatinine clearance more than 60 ml / min)

Normal liver function (AST, ALT - no more than 3 norms)

Left ventricular ejection fraction> 55%

Adequate marrow function (hemoglobin level more than 9 g / dL, neutrophil count more than 1.5 thousand / μl, platelet number more than 100 thousand / μl)

Signed informed consent

Exclusion Criteria:

Children, women during pregnancy, childbirth, women during breastfeeding

Persons with mental disorders

The presence of an active viral infection with HIV, viral hepatitis B and C

Inoperable tumor

Morphologically confirmed diagnosis of GIST, Kaposi's sarcoma, alveolar or clear cell sarcoma, chondrosarcoma, chordoma, giant cell tumor, paraosal osteosarcoma, Ewing's sarcoma / PNET, rhabdomyosarcoma, G1 osteosarcoma

The presence of a second malignant neoplasm within the last 5 years before enrollment, other than cured basal cell or squamous cell carcinoma or cervical cancer in situ, prostate cancer

Clinically significant cardiovascular or cerebrovascular diseases within the last 6 months (acute myocardial infarction, unstable angina pectoris, significant ventricular arrhythmias, severe heart failure (NYHA class IV), stroke or uncontrolled arterial hypertension)

Renal failure (serum creatinine level more than 150 μmol / L), except for cases caused by lymphoid infiltration of the kidneys, and tumor disintegration syndrome

Hepatic failure (except for cases caused by leukemic / lymphoid organ infiltration), acute hepatitis (serum bilirubin level more than 2 norms, ALT and AST activity more than 4 norms, prothrombin index less than 50%)

Decompensated diabetes mellitus (blood serum glucose above 15 mmol / L)

Sepsis (septicopyemic foci, hemodynamic instability; ineffective antimicrobial therapy) or acute infectious diseases

Brain metastases

Life-threatening conditions (bleeding, tumor decay, etc.)

Hypersensitivity to the active substance of the investigational drugs or any of the auxiliary components or their intolerance

Surgical interventions less than 21 days before starting therapy

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months
  Proportion of patients who have a partial or complete response to therapy

SECONDARY OUTCOMES:
Comparison of tumor necrosis | 6 months
  Proportion of tumor necrosis after chemotherapy
Comparison of safety assessment | 6 months
  Adverse Event Assessment and Serious Adverse Event Assessment according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Beniamin Bokhyan, PhD, Principal Investigator — N.N. Blokhin NMRCO
Locations (1):
- Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" оf the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official site — https://www.ronc.ru/about/struktura/niiko/ooo/hn1/
- See also: russian surcoma group site — https://sarcomarus.ru/